CLINICAL TRIAL: NCT03288181
Title: Effects of Muscle Stretching on Vascular Endothelial Function in Patients With Peripheral Arterial Disease
Brief Title: Effects of Passive Muscle Stretching on Vascular Function and Symptoms of PAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tallahassee Research Institute, Inc. (Other)
Collaborators: Florida State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2015-25
Record Dates: First submitted 2017-09-15; First posted 2017-09-19 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Peripheral Arterial Disease; Claudication
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle Stretch Group (Experimental): This is the group who applies the splint to stretch the calf muscles as per the described protocol for 4 weeks.
  Interventions: Device: Muscle Stretch
- Control Arm (No Intervention): This is the group who has undergone no splint for 4 weeks.

INTERVENTIONS:
Device: Muscle Stretch — The splint will be applied to the affected leg as per the protocol for 30 minutes per day, 5 days per week for 4 weeks.
  Arms: Muscle Stretch Group

SUMMARY:
Patients with peripheral arterial disease often have walking impairment due to insufficient oxygen supply to lower extremity skeletal muscle. In an aging rat model, we have previously shown that daily calf muscle stretching improves endothelium-dependent dilation of soleus muscle arterioles and blood flow during exercise. The effect of muscle stretching on endothelial function and walking distance in patients with peripheral arterial disease is unknown. We performed a prospective, randomized, non-blinded, crossover study in 13 patients with stable symptomatic peripheral artery disease. Patients were randomized to undergo either 4 weeks of passive calf muscle stretching (ankle dorsiflexion splints applied 30 minutes/day, 5 days/week) followed by 4 weeks of no muscle stretching (control group) and vice versa. Endothelium-dependent flow-mediated dilation and endothelium- independent nitroglycerin-induced dilation of the popliteal artery and a 6 minute walk test were evaluated at baseline and after each 4 week treatment interval. Patients crossed over to the other treatment arm after 4 weeks and endothelium-dependent flow-mediated dilation and endothelium- independent nitroglycerin-induced dilation of the popliteal artery and the 6 minute walk test were repeated.

DETAILED DESCRIPTION:
This study is a prospective randomized, non-blinded, crossover trial conducted at Tallahassee Memorial HealthCare, Tallahassee, FL, USA between October 2015 and May 2016. The Tallahassee Memorial Healthcare Institutional Review Board and the Human Subject Committee at Florida State University approved the study prior to initiation. Informed written consent was provided by all patients prior to enrollment.

Study Patients The study sample consisted of patients with stable symptomatic PAD. Inclusion criteria included reproducible claudication with walking associated with an ankle brachial index of less than 0.90,15 and/or computed tomographic angiographic evidence of at least a 60% stenosis of the iliac, femoral, or popliteal artery deemed to be the source of claudication. Individuals with critical limb ischemia or who had severe comorbid conditions limiting their walking ability were excluded.

Study Design:

Participants were initially randomized to undergo either 4 weeks of passive stretching or 4 weeks of no stretching (control), respectively, followed by cross-over to the other intervention. Patients were evaluated at baseline, after the first 4 weeks of initial intervention (stretching or no stretching) and then again after 4wks following the cross-over intervention (stretching or no stretching). Participants were taught how to apply a simple dorsiflexion splint and during the 4 wks of daily stretching intervention and applied the splint daily at home for 30 minutes/day, 5 days/week. Endothelium-dependent flow-mediated dilation (FMD) and endothelium-independent nitroglycerin-induced dilation (NID) of the popliteal artery (measured by doppler ultrasound) and a 6 minute walk test were evaluated at baseline and after each 4 week treatment interval.

Muscle stretching Protocol. To passively stretch each patient's calf muscle, dorsiflexion splints (Healwell Plantar Fasciitis Night Splint®, FLA Orthopedics, Charlotte, NC, USA) were applied. Using the splint, ankle joints were kept at 15 degrees of dorsiflexion for 30 min/day, 5 days/wk, for the 4 week interval. The splint has a strap to adjust the angle of the joint. Participants learned how to wear the splint correctly from a trained physical therapist who initially fitted and adjusted the splint. Splints were sent home with the patient and a physical therapist was available for questions by phone. Using the splint, both the gastrocnemius and soleus muscles were effectively stretched. If participants complained of pain during muscle stretching, the physical therapist assisted in adjusting the straps, but efforts were made to maintain the angle of dorsiflexion.

Flow-mediated dilation of the popliteal artery. Vascular functional testing was performed in a temperature controlled (72 degrees F), quiet and dark laboratory. To exclude the acute effects of acute exercise or medicine on vascular endothelial function, participants were asked to refrain from taking sildenafil, tadalafil and vardenafil for 48 hours prior to the vascular assessment, and not to take carvedilol, cartelol labetalol, verapamil, diltiazem, nifedipine, nicardipine, isradipine, felodipine and amlodipine for 24 hours prior to the assessment. Participants were also asked to refrain from any form of exercise and not to eat or drink for 3 hours prior to the assessment.

Systolic and diastolic blood pressure was measured using an automatic brachial sphygmomanometer applied to the upper arm after at least 10 min of quiet rest with the patient seated in the vascular laboratory. Pulse rate was recorded. Participants then assumed a prone position on a bed and a blood pressure cuff applied to the lower thigh of the most symptomatic lower extremity. Using vascular ultrasound and Doppler (GE Vivid Q ultrasound with 12L-RS Linear Vascular Probe, GE, Milwaukee, WI, USA), flow-mediated dilation of the popliteal artery was measured in the following manner. The measurement was conducted on the affected leg (leg with greater symptoms or lower ankle-brachial index). First, popliteal artery diameter and blood flow velocity were recorded after resting for 10 min. A lower thigh blood pressure cuff was then inflated up to 250 mmHg for 5 min. During the 5 min of arterial occlusion, participants were asked to remain as still as possible. The blood pressure cuff was then quickly deflated, and popliteal artery diameter and blood flow remeasured in the same location for another 10 min. FMD was obtained by referencing the peak popliteal artery diameter to the baseline measurement.

Endothelium-independent dilation of the popliteal artery. At least 30 min after the assessment of FMD, nitroglycerin-induced dilation (NID) of the popliteal artery was also assessed as a measure of endothelium-independent dilation. Baseline popliteal artery diameter was recorded after resting for 10 min. The recording was done continuously for 10 min after the administration of 400 µg of sublingual nitroglycerin (NTG, Wilshire, Atlanta, Georgia). The peak diameter relative to baseline served as the measurement of endothelium-independent dilatation.

Hemodynamic analyses. Vessel diameter and blood flow velocity were recorded at 30 Hz of frequency, and converted into DICOM (DICOM, Rosslyn, VA, USA) format to perform further analysis. Since peripheral arterial diameter and blood flow velocity vary during the cardiac cycle,16 popliteal artery diameter was measured at the end of the diastolic phase (defined as the point just before the popliteal arterial Doppler waveform rises). Blood flow velocity was measured at the peak of the systolic phase. Using two-dimensional B mode images, end-diastolic popliteal artery diameter and peak velocity were obtained from three consecutive cardiac cycles, averaged and the same technique used to measure arterial diameter for FMD and NID.

Six-minute Walk Test (6MWT) The Six-minute walk test (6MWT) was performed after vascular function testing according to the American Thoracic Society guidelines.Using a straight 30m corridor, participants were asked to walk back and forth over 6 minutes. Participants were asked to report any symptoms, including leg pain or cramping, tiredness and/or chest discomfort. Participants were allowed to rest if they felt it necessary and then asked to resume walking as soon as able. Symptom-free walking distance was measured as the distance covered without symptoms. Continuous walking distance was also measured as the distance covered without stopping. Total 6-minute walking distance was measured as the distance covered for 6 minutes. Immediately after the 6-minute walk, participants were seated and again asked to report any chest and lower-extremity symptoms. Chest and lower-extremity exertional symptoms were assessed using a modified borg scale. The modified borg scale is scored from zero (no symptoms of exertion) to 10 (maximal sensation of symptoms). Participants answered the chest and lower-extremity symptoms by indicating a number from zero to 10. Systolic and diastolic blood pressure and heart rate were then measured at approximately 1-min after 6-min walk termination.

Sample size calculation. The primary endpoint for which the sample size was derived was popliteal artery FMD. From published data, we estimated that the FMD of popliteal artery would improve by approximately 40% with muscle stretching. In a prior pilot study, we observed a baseline FMD of 3.87% (standard deviation of 0.62%) in 13 patients with stable PAD. Assuming an alpha of 0.05, and a cross-over design, we predicted that we would need at least 12 patients per group to have 90% power to detect a 20% increase in FMD. Allowing for an approximately 20% drop out rate (3 patients), the targeted sample size was adjusted to 15 in this study. However, recruitment was to continue until at least 12 patients were enrolled and completed the protocol.

Statistical analysis. Baseline clinical characteristics are reported as means and standard deviations. A histogram of vascular function and walking distance was made to assess their distribution. If non-normal distribution was suggested by the histogram, a Kolmogorov-smirnov test was performed to assess the distribution of obtained data. On the basis of the distribution test, paired t-test (normal distribution) or Wilcoxon signed-rank test (non-normal distribution) were used to compare between those data obtained after 4 weeks of stretching and after 4 weeks of no stretching with a 2-sided level of significance of 0.05. Data were presented as mean ± standard error.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable symptomatic peripheral arterial disease

Exclusion Criteria:

* critical limb ischemia
* severe comorbid conditions that limit walking ability

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-10-05 (Actual); Primary Completion 2016-05-30 (Actual); Study Completion 2016-06-15 (Actual)

PRIMARY OUTCOMES:
Flow Mediated Dilatation of the Popliteal Artery | Performed 4 weeks after each intervention
  Ultrasound assessment of flow mediated dilatation of the popliteal artery

SECONDARY OUTCOMES:
Six Minute Walk Test | Performed 4 weeks after each intervention
  Standard 6 minute walk test to evaluate walking distance

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Batchelor, MD, Principal Investigator — Tallahassee Research Institute

IPD SHARING:
Plan to Share IPD: No